CLINICAL TRIAL: NCT07305454
Title: Impact of a Structured Therapeutic Education Session on the Practice of Adapted Physical Activity in Chronic Inflammatory Bowel Diseases
Acronym: ETAP-MICI
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/25/0588; ID-RCB (Other: 2025-A02645-44)
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Chronic Inflammatory Bowel Disease
Keywords: chronic inflammatory bowel disease; crohn disease; ulcerative colitis; physical activity
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with chronic inflammatory bowel disease: patients with chronic inflammatory bowel disease in clinical remission
  Interventions: Diagnostic Test: Inflammatory Bowek Disk Questionnaires; Other: Short-International Physical Activity Questionnaries

INTERVENTIONS:
Diagnostic Test: Inflammatory Bowek Disk Questionnaires — Patients will be asked to complete the questionnaires regarding bowel inflammation at enrollment, 6 months later, and 12 months later.
Other: Short-International Physical Activity Questionnaries — Patients will be asked to complete the physical activity questionnaire 6 months later and 12 months later.

SUMMARY:
Chronic inflammatory bowel diseases (IBD; including Crohn's disease and ulcerative colitis) significantly impact patients' quality of life. Among non-pharmacological therapies, adapted physical activity (APA) has demonstrated its beneficial impact, particularly on fatigue, anxiety, digestive symptoms, and the overall quality of life of patients with IBD.

The real-world implementation of APA remains insufficient, primarily due to limited patient adherence to this prescription.

Patient therapeutic education (PTE) represents a potentially powerful lever for promoting engagement in APA by addressing barriers related to a lack of awareness (fear of symptom worsening) and lack of motivation. No dedicated study has specifically evaluated the effect of targeted PTE sessions on adherence to physical activity in IBD.

The objective of our feasibility study will be to determine whether a single therapeutic education session focused on the digestive and systemic benefits of APA has an impact on the rate of physical activity practice in the medium term among patients with IBD in clinical remission for at least 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Inflammatory Bowel Disease
* Age > 18 years
* Crohn's disease in clinical remission (defined by a Harvey Bradshaw Index ≤ 5) or ulcerative colitis in clinical remission (defined by a Mayo score < 3 and no subscore > 1) for at least 3 months
* Social Security coverage

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Patient under legal guardianship
* Cardiovascular or rheumatic conditions contraindicating participation in sports
* Neurological conditions with residual deficits contraindicating participation in sports
* Refusal or inability to consent to participation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic inflammatory bowel disease in clinical remission (Crohn's disease or ulcerative colitis)
Sampling Method: Non-Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of therapeutic education intervention on physical activity practice | 12 months after the inclusion
  Measure the amount of metabolic equivalent or MET/Week (Metabolic Equivalent Task) at 12 months, based on the short-IPAQ questionnaire assessing physical activities reported by the patient over the last 7 days.

SECONDARY OUTCOMES:
study the impact on quality of life at 6 months | 6 months after the inclusion
  measure of quality of life with the IBD disk questionnaires answers at 6 months
Study the impact on quality of life in 12 months | 12 months after the inclusion
  measure of quality of life with the IBD disk questionnaires answers at 12 months
study the impact on fatigue reported at 6 months | 6 months after the inclusion
  Measure of fatigue reported according to one of the items of the IBD Disk questionnaire at 6 months
study the impact on fatigue reported at 12 months | 12 months after the inclusion
  Measure of fatigue reported according to one of the items of the IBD Disk questionnaire at 12 months
study the correlation between increased overall muscle strength and improved quality of life | 12 months after the inclusion
  Measurement of estimated muscle strength using a hand grip test before and after intervention as part of annual malnutrition screening and response to the quality of life questionnaire
Study of the impact on the evolution of IBD activity at 6 months | 6 months after the inclusion
  measurement of clinical activity in chronic inflammatory bowel disease at 6 months
Study of the impact on the evolution of IBD activity at 12 months | 12 months after the inclusion
  measurement of clinical activity in chronic inflammatory bowel disease at 12 months
study the impact on the monitoring of the prescription of adapted physical activity | 12 months after the inclusion
  Monitoring of the APA prescription estimated according to the proportion of patients who completed at least 12 APA sessions (i.e. 1 weekly session for 3 months) and the average number of APA sessions completed.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gastro-Entérologie, CHU Toulouse, Hôpital Rangueil, 1 avenue Jean Poulhès, Toulouse, France

IPD SHARING:
Plan to Share IPD: No